CLINICAL TRIAL: NCT07056465
Title: Acceptability of, and Compliance to a Novel Intermittent Carbohydrate Restriction Dietary Intervention
Brief Title: Exploring Adherence and Acceptability of an Intermittent Carbohydrate Restriction Regime in Free-Living Adults: A Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FHMS 22-23 054 EGA
Record Dates: First submitted 2025-06-05; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Healthy
Keywords: intermittent carbohydrate restriction; feasibility study; dietary intervention; Behavioural change; Body composition
MeSH Terms: interventions — Clinical Protocols

STUDY DESIGN:
Intervention Model Description: single-arm feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-Arm Intermittent Carbohydrate Restriction Intervention (Experimental): Participants in this single-arm feasibility study will follow a structured intermittent carbohydrate restriction (ICR) dietary protocol for four weeks. The ICR approach includes two non-consecutive low-carbohydrate days (≤40g/day) and five habitual eating days per week. The intervention is designed to assess dietary adherence, acceptability, and impact on body composition and food preferences in free-living healthy adults. Data will be collected through anthropometric measurements, dietary assessments (food diaries and 24-hour recalls), and participant-reported outcomes via questionnaires and exit interviews.
  Interventions: Behavioral: Intermittent Carbohydrate Restriction (ICR) Protocol

INTERVENTIONS:
Behavioral: Intermittent Carbohydrate Restriction (ICR) Protocol — A novel intermittent carbohydrate restriction (ICR) protocol involving two consecutive low-carbohydrate days (approximately 10% total energy from carbohydrate) followed by five non-restricted days per week, sustained over a 4-week period. Participants receive individualised dietary guidance and support materials to promote adherence in free-living conditions

SUMMARY:
This study investigates a novel dietary approach called Intermittent Carbohydrate Restriction (ICR), which involves reducing carbohydrate intake on selected days of the week while allowing habitual eating on other days. Previous research suggests that intermittent dietary strategies may improve metabolic health and support better adherence compared to continuous calorie restriction.

In this single-arm feasibility study, 40 healthy adults will follow the ICR protocol for 4 weeks. Outcomes including body weight, body fat percentage, waist circumference, and resting metabolic rate will be measured before and after the intervention. Dietary adherence, changes in habitual intake, and participant experiences will be assessed through food diaries, 24-hour recalls, questionnaires, and exit interviews.

The primary aim is to evaluate the acceptability and adherence to the ICR protocol in free-living conditions. Secondary aims include exploring its effects on body composition and diet-related behaviours, with the goal of informing future long-term dietary interventions.

DETAILED DESCRIPTION:
Intermittent energy restriction (IER) has shown to improve postprandial metabolic systems and cognitive function, with superiority in dietary adherence compared with continuous energy restriction (CER)(1-3). A gap in current research is the impact of intermittent carbohydrate restriction (ICR) compared with IER in line with the carbohydrate-insulin model. Novel research (UEC 2019 008 FHMS) has explored the acute effects of ICR on postprandial metabolic systems and found engagement of the same underlying mechanisms with superior outcomes in glucose and lipid metabolism, compared with IER. Unpublished data supports the superiority of ICR over IER in dietary adherence due to perceived increased flexibility and reduced restrictions. However, a novel intermittent carbohydrate restricted diet has not been studied chronically, specifically exploring effects adherence and compliance on free living condition and its effect on body composition and food preference. This study primarily aims to explore the acceptability and compliance to ICR, and secondarily aims to explore its effect on behaviour change and body composition in free living condition in health adults. 40 participants (female and male) will follow a single arm novel intermittent carbohydrate diet protocol for 4 weeks. Weight, height, body fat %, waist circumference and resting energy expenditure values will be measured before and after the intervention. Compliance and the effects of dieting on the habitual food intake will be measured using food diaries and 24hr food recalls. Perceptions of participants' towards ICR and their experiences of dieting will be measured using questionnaires and an exit interview. This study will provide vital information for implementing flexible and adaptable dieting strategy, which can provide improvements to physical health in the long-term.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 18.5 and 29.9 kg/m² (normal to overweight range; avoids confounding from obesity-related metabolic disturbances).
* Generally healthy (self-reported good health with no diagnosed metabolic, cardiovascular, or endocrine disorders).
* Not currently following a weight-loss diet or carbohydrate-restricted diet (to ensure dietary baseline is not already influenced by similar patterns).
* Willing and able to follow the ICR protocol for 4 weeks (includes ability to prepare meals and follow dietary instructions independently).
* Able to attend in-person laboratory assessments at baseline and follow-up (for measurements of REE, body composition, etc.).
* Fluent in English (to ensure comprehension of dietary instructions, consent forms, and interviews).
* Provides written informed consent (as per ethical standards and good clinical practice).

Exclusion Criteria:

* Diagnosed metabolic or endocrine disorders (e.g., diabetes, hypothyroidism, PCOS), to avoid confounding effects on metabolic outcomes and dietary adherence.
* History of cardiovascular disease, renal disease, or gastrointestinal disorders (e.g., IBS, coeliac disease), which may affect dietary tolerance or nutrient absorption.
* Currently pregnant, breastfeeding, or planning pregnancy during the study (due to potential risks and altered metabolic/nutritional needs).
* BMI <18.5 or ≥30 kg/m² (to exclude underweight or obese individuals where safety and generalizability may differ).
* Currently following a restrictive or structured diet (e.g., ketogenic, low-carb, intermittent fasting, or weight-loss diets), to ensure a clear baseline dietary behavior.
* History or presence of eating disorders (e.g., anorexia nervosa, bulimia, binge eating), for participant safety and ethical considerations.
* Use of medications or supplements known to affect metabolism or appetite (e.g., corticosteroids, GLP-1 agonists, weight-loss medications).
* Smoking or excessive alcohol consumption (defined as >14 units/week), which may interfere with dietary adherence and metabolic assessments.
* Participation in another clinical or dietary study within the past 3 months (to avoid overlapping interventions or residual effects).
* Inability or unwillingness to comply with study procedures (including dietary tracking, visit attendance, or sample collection).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2023-01-13 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-04-20 (Actual)

PRIMARY OUTCOMES:
Adherence to the ICR protocol | Throughout the 4-week intervention
  Assessed quantitatively as the proportion of participants who successfully follow the prescribed dietary regimen (≥75% of prescribed LC-Ds completed over 4 weeks), measured through 24-hour recalls.

SECONDARY OUTCOMES:
Change in body weight (kg) | Baseline (Week 1) and Week 4 (Final study day)
  Measured before and after the 4-week intervention using standard anthropometric techniques.
Changes in resting energy expenditure (kcal/day) | Baseline (Week 1) and Week 4 (Final study day)
  Assessed via indirect calorimetry before and after the intervention. Includes respiratory quotient (RQ) as a metabolic indicator.
Change in daily energy intake (kcal/day) | Baseline (Week 1) and Week 4 (Final study day)
  Assessed via food diaries and 24-hour dietary recalls.
Participant experiences with the ICR intervention (qualitative interview) | Week 4 (final study day)
  Exploratory assessment of participants' behavioral and psychological responses to the ICR intervention, including perceived changes in food preferences and attitudes toward carbohydrate-containing foods . Data will be collected via semi-structured exit interviews and analysed using thematic analysis.
Change in body fat percentage (%) | Baseline (Week 1) and Week 4 (Final study day)
  Measured before and after the 4-week intervention using [method, e.g., bioelectrical impedance
Change in waist circumference (cm) | Baseline (Week 1) and Week 4 (Final study day)
  Measured before and after the 4-week intervention at the midpoint between the iliac crest and lowest rib.
Change in respiratory quotient (VCO₂/VO₂) | Baseline (Week 1) and Week 4 (Final study day)
  Assessed via indirect calorimetry before and after the intervention.
Change in macronutrient distribution (% total energy intake) | Throughout the 4-week intervention
  Assessed via food diaries and 24-hour dietary recalls.
Change in micronutrient distribution (% total energy intake) | Throughout the 4-week intervention
  Assessed via food diaries and 24-hour dietary recalls.
Change in vegetable intake (servings/day) | Throughout the 4-week intervention
  Assessed via food diaries and 24-hour dietary recalls.
Change in oily fish intake (g/week) | Throughout the 4-week intervention
  Assessed via food diaries and 24-hour dietary recalls.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Wells, Dr, Study Chair — University of Surrey
Locations (1):
- University of Surrey, Guildford, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Biyikoglu H, Robertson MD, Collins AL. Isolating the acute metabolic effects of carbohydrate restriction on postprandial metabolism with or without energy restriction: a crossover study. Eur J Nutr. 2025 Mar 20;64(3):133. doi: 10.1007/s00394-025-03646-5. PMID 40111529
- [Derived] Biyikoglu H, Tse YT, Ding R, Mold FE, Collins AL. Exploring Adherence and Acceptability of an Intermittent Carbohydrate Restriction Regime (ICARB) in Free-Living Adults: A Feasibility Study. J Hum Nutr Diet. 2026 Feb;39(1):e70188. doi: 10.1111/jhn.70188. PMID 41536043